CLINICAL TRIAL: NCT02158468
Title: Effect of Conditioning on Myocardial Damage in ST-elevation Myocardial Infarction - Comparison of Combined Intrahospital Preconditioning Plus Postconditioning Versus Postconditioning Versus Control.
Brief Title: Effect of Conditioning on Myocardial Damage in STEMI
Acronym: LIPSIA-COND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIPSIA-Conditioning
Record Dates: First submitted 2014-05-26; First posted 2014-06-06 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2014-12

CONDITIONS: ST-elevation Myocardial Infarction
Keywords: STEMI, reperfusion, preconditioning, postconditioning, reperfusion injury, myocardial salvage
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Reperfusion Injury | interventions — Ischemic Postconditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Combined intrahospital pre- and postconditioning (Active Comparator): After admission to hospital 3 cycles of preconditioning with 5-min inflation and 5-min deflation of a blood-pressure cuff. After primary PCI/stenting 4 cycles of postconditioning (30s ischemia and 30s reperfusion).
  Interventions: Device: Combined intrahospital pre- and postconditioning
- Postconditioning (Active Comparator): 4 cycles of postconditioning (30s ischemia, 30s reperfusion) after primary PCI/stenting
  Interventions: Device: Postconditioning
- Control group (No Intervention): Standard infarction treatment without conditioning intervention

INTERVENTIONS:
Device: Combined intrahospital pre- and postconditioning — After admission to hospital 3 cycles of preconditioning with 5-min inflation and 5-min deflation of a blood-pressure cuff. After primary PCI/stenting 4 cycles of postconditioning (30s ischemia and 30s reperfusion)
  Arms: Combined intrahospital pre- and postconditioning
Device: Postconditioning — After primary PCI/stenting 4 cycles of postconditioning (30s ischemia and 30s reperfusion)
  Arms: Postconditioning

SUMMARY:
The LIPSIA-Conditioning trial is an investigater initiated, randomized, single-center study that will assess the effect of different intrahospital conditioning protocols on myocardial damage assessed by MRI in patients with acute ST-elevation myocardial infarction.

The following groups will be compared:

1. Combined intrahospital pre- plus postconditioning versus
2. Postconditioning versus
3. Control

DETAILED DESCRIPTION:
Rapid reperfusion of the infarct-related coronary artery is essential to salvage ischemic myocardium in patients with acute ST-elevation myocardial infarction (STEMI). Paradoxically, restoration of the blood flow to the ischemic area may result in further injury to the myocardium.

This phenomenon is described as 'ischemia/reperfusion injury' and the pathophysiological mechanisms are not fully elucidated. A cardioprotective effect of ischemic preconditioning as well for postconditioning (short repetitive cycles of reperfusion and re-occlusion) has been demonstrated in experimental studies and in pilot studies on patients with acute STEMI treated with primary percutaneous coronary intervention.

Aim of this study is to compare for the first time the combination of intrahospital pre- and postconditioning versus exclusive postconditioning versus control. The primary endpoint of this study will be the salvaged area at risk assessed by cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

ST-elevation myocardial infarction <12 hours

Exclusion Criteria:

* Age ≤ 18 years
* Patients presenting with pregnancy
* Thrombolysis <12 hours
* Patients without informed consent
* Participation in another trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2011-10; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage assessed by MRI | 1 week after infarction

SECONDARY OUTCOMES:
Composite of death, reinfarction and readmission for congestive heart failure | 6 months

OTHER OUTCOMES:
Infarct size assessed by MRI | 1 week after infarction
Microvascular obstruction assessed by MRI | 1 week after infarction

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Eitel, MD, Principal Investigator — University Leipzig- Heart Center
Locations (1):
- University Leipzig - Heart Center, Department of Cardiology, Leipzig, Please Select, Germany

REFERENCES:
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Lonborg J, Kelbaek H, Vejlstrup N, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Treiman M, Jensen JS, Engstrom T. Cardioprotective effects of ischemic postconditioning in patients treated with primary percutaneous coronary intervention, evaluated by magnetic resonance. Circ Cardiovasc Interv. 2010 Feb 1;3(1):34-41. doi: 10.1161/CIRCINTERVENTIONS.109.905521. Epub 2010 Jan 26. PMID 20118154
- [Derived] Lange T, Gertz RJ, Schulz A, Backhaus SJ, Evertz R, Kowallick JT, Hasenfuss G, Desch S, Thiele H, Stiermaier T, Eitel I, Schuster A. Impact of myocardial deformation on risk prediction in patients following acute myocardial infarction. Front Cardiovasc Med. 2023 Aug 10;10:1199936. doi: 10.3389/fcvm.2023.1199936. eCollection 2023. PMID 37636296
- [Derived] Stiermaier T, Jensen JO, Rommel KP, de Waha-Thiele S, Fuernau G, Desch S, Thiele H, Eitel I. Combined Intrahospital Remote Ischemic Perconditioning and Postconditioning Improves Clinical Outcome in ST-Elevation Myocardial Infarction. Circ Res. 2019 May 10;124(10):1482-1491. doi: 10.1161/CIRCRESAHA.118.314500. PMID 30929570
- [Derived] Saad M, Stiermaier T, Fuernau G, Poss J, de Waha-Thiele S, Desch S, Thiele H, Eitel I. Impact of direct stenting on myocardial injury assessed by cardiac magnetic resonance imaging and prognosis in ST-elevation myocardial infarction. Int J Cardiol. 2019 May 15;283:88-92. doi: 10.1016/j.ijcard.2018.11.141. Epub 2018 Dec 3. PMID 30573280
- [Derived] Stiermaier T, Jobs A, de Waha S, Fuernau G, Poss J, Desch S, Thiele H, Eitel I. Optimized Prognosis Assessment in ST-Segment-Elevation Myocardial Infarction Using a Cardiac Magnetic Resonance Imaging Risk Score. Circ Cardiovasc Imaging. 2017 Nov;10(11):e006774. doi: 10.1161/CIRCIMAGING.117.006774. PMID 29122844
- [Derived] Reinstadler SJ, Stiermaier T, Liebetrau J, Fuernau G, Eitel C, de Waha S, Desch S, Reil JC, Poss J, Metzler B, Lucke C, Gutberlet M, Schuler G, Thiele H, Eitel I. Prognostic Significance of Remote Myocardium Alterations Assessed by Quantitative Noncontrast T1 Mapping in ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Imaging. 2018 Mar;11(3):411-419. doi: 10.1016/j.jcmg.2017.03.015. Epub 2017 Jun 14. PMID 28624398
- [Derived] Eitel I, Stiermaier T, Rommel KP, Fuernau G, Sandri M, Mangner N, Linke A, Erbs S, Lurz P, Boudriot E, Mende M, Desch S, Schuler G, Thiele H. Cardioprotection by combined intrahospital remote ischaemic perconditioning and postconditioning in ST-elevation myocardial infarction: the randomized LIPSIA CONDITIONING trial. Eur Heart J. 2015 Nov 21;36(44):3049-57. doi: 10.1093/eurheartj/ehv463. Epub 2015 Sep 17. PMID 26385956